CLINICAL TRIAL: NCT00870584
Title: A 26-week Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Effect of Omalizumab on Markers of Asthma Impairment in Patients With Persistent Allergic Asthma
Brief Title: Evaluate the Effect of Omalizumab on Markers of Asthma Impairment in Patients With Persistent Allergic Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025AUS33
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Results first posted 2011-11-17 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-10

CONDITIONS: Persistent Allergic Asthma
Keywords: Asthma; asthma management; asthma impairment ; Xolair ; omalizumab
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Omalizumab (Experimental): The determined dose (at least 0.016 mg/kg/IgE (IU/mL) was administered subcutaneously every 2 weeks or every 4 weeks. Dose and dosing interval were determined based on patient body weight and pre-treatment serum IgE level; a dosing table was used.
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): Placebo was administered subcutaneously every 2 weeks or every 4 weeks depending on the dosing schedule in the protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — Omalizumab was supplied as a lyophilized, sterile powder in a single-use, 5 mL vial. The vial was designed to deliver 150 mg (1.2 mL) of omalizumab for subcutaneous (s.c.) administration after reconstitution with 1.4 mL sterile water for injection. Doses of more than 150 mg were divided among multiple injection sites to limit injections to not more than 150 mg per site.
  Other Names: Xolair
  Arms: Omalizumab
Drug: Placebo — Placebo was supplied as a lyophilized, sterile powder in a single-use, 5 mL vial. The vial was designed to deliver 150 mg (1.2 mL) of placebo for subcutaneous (s.c.) administration after reconstitution with 1.4 mL sterile water for injection. Doses of more than 150 mg were divided among multiple injection sites to limit injections to not more than 150 mg per site.
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of omalizumab on markers of impairment in patients with inadequately controlled persistent allergic asthma on Step 4 or above therapy as defined in the 2007 National Heart, Lung, and Blood Institute (NHBLI) Guidelines

ELIGIBILITY:
Inclusion Criteria:

* Total Asthma Control Test (ACT) score of ≤19 plus at least one of the following in the 4 weeks preceding visit 1, on average:

  * Symptoms > 2 days/week
  * Night-time awakenings ≥1 time/week
  * Short-acting beta2-agonist (SABA) use for symptom control >2 days/week forced expiratory volume in 1 second (FEV1) ≤ 80% predicted

Exclusion Criteria:

* History of intubation for asthma.
* An asthma exacerbation requiring treatment with systemic steroids within 4 weeks of screening (Visit 1).
* Less than 3 months of stable maintenance oral corticosteroid therapy for asthma

Other protocol-defined inclusion/exclusion criteria applied

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (50):
- United States (50):
  - Jasper Summit Research, LLC, Jasper, Alabama
  - Allergy Asthma and Immunology Center of Alaska, Anchorage, Alaska
  - Medical Research of Arizona, A division of Allergy Asthma & Immunology Associates, LTD, Scottsdale, Arizona
  - Waren W. Pleskow, MD, Encinitas, California
  - William Ebbeling, MD, Inc, Fresno, California
  - Pediatric Care Medical Group, Inc, Huntington Beach, California
  - California Allergy & Asthma Medical Group, Palmdale, California
  - Allergy Associates Medical Group, Inc, San Diego, California
  - Sansum Clinic, Santa Barbara, California
  - Allergy & Asthma Clinical Research, Inc., Walnut Creek, California
  - Innovative Research of West Florida, Inc, Clearwater, Florida
  - Palm Spring Research Institute, Inc, Hialeah, Florida
  - Integrity Research, LLC, Pensacola, Florida
  - Hugh Windom, MD, PA, Sarasota, Florida
  - South Miami Clinical Research, LLC, South Miami, Florida
  - Georgia Pollens Clinical Research Centers, Inc, Albany, Georgia
  - Sneeze, Wheeze and Itch Associates, LLC, Normal, Illinois
  - Chest Medicine Clinical Services, Skokie, Illinois
  - Clinical Research Center of Indiana, Indianapolis, Indiana
  - Kansas City Allergy & Asthma Center, Overland Park, Kansas
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - Abraham Research, PLLC, Crescent Springs, Kentucky
  - Rx R&D, Metairie, Louisiana
  - Acadiana Medicine Clinic, Opelousas, Louisiana
  - Paul A Shapero, MD, Bangor, Maine
  - Chesapeake Clinical Research, Baltimore, Maryland
  - Respiratory Medicine Research Institute of Michigan, Ypsilanti, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - Maimonides Medical Center, Division of Pediatric Pulmonology, Brooklyn, New York
  - Allergy Asthma Immunology of Rochester Research Center, Rochester, New York
  - Alan Kaufman, MD, The Bronx, New York
  - Allergy & Asthma Center of NC, PA, High Point, North Carolina
  - Wilmington Medical Research, Wilmington, North Carolina
  - Allergy and Respiratory Center, Canton, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Oklahoma Allergy & Asthma Clinic, Oklahoma City, Oklahoma
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Baker Allergy Asthma and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Asthma Allergy & Pulmonary Associates, Philadelphia, Pennsylvania
  - AAPRI Clinical Research Institute, Lincoln, Rhode Island
  - Pediatric Pulmonary Associates of North Texas, PA, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - North Texas Institute for Clinical Trials, Fort Worth, Texas
  - Allergy & Asthma Associates, Houston, Texas
  - Lynchburg Pulmonary Associates, Lynchburg, Virginia
  - Virginia Adult and Pediatric Allergy and Asthma PC, Richmond, Virginia
  - Asthma Inc., Seattle, Washington
  - Pulmonary and Research Associates, Spokane, Washington

REFERENCES:
- See also: Related Info — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 136 | 135
Completed | 120 | 122
Not Completed | 16 | 13
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Lost to Follow-up | 5 | 1
Not completed — Protocol Deviation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 136 | 135 | 271
Age Continuous [Mean (Standard Deviation); unit: years] | 41.9 (14.60) | 40.7 (14.85) | 41.3 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 87 | 180
  Male | 43 | 48 | 91

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Asthma Control Test (ACT) After 24 Weeks of Treatment
Description: The Asthma Control Test (ACT) is a validated tool to assess overall asthma control over the last 4 weeks in patients aged >= 12 years old. It is a 1 page questionnaire consisting of 5 simple questions assessing: asthma symptoms, use of rescue medications, and the impact of asthma on everyday functioning. All questions are scored on a 5-point Likert scale, with a higher score indicating better control. All scores are added together to calculate a total score. Total score ranges from 5 to 25. A positive change indicates improvement.
Time Frame: Baseline and 24 weeks
Population: The Full Analysis Set consisted of patients to whom study drug had been assigned through randomization. Patients inappropriately randomized were excluded from this analysis set.
  Participants with observations at both baseline and 24 weeks were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 118 | 123
Score on a scale | 5.2 (4.37) | 4.7 (4.01)

2. Secondary Outcome: Investigator Global Evaluation of Treatment Effectiveness (IGETE) at 24 Weeks
Description: The IGETE is an assessment of asthma symptom control in response to asthma treatment. It consists of the question "What is the investigator's overall impression of the study medication and its effect on the typical symptoms of allergic asthma during the study?" The scale is: excellent, good, moderate, poor, and worsening. A good or excellent response is suggested as a means of defining a patient who has responded to treatment.
Time Frame: 24 weeks
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 136 | 135
participants
  Excellent | 26 | 19
  Good | 44 | 44
  Moderate | 29 | 30
  Poor | 27 | 36
  Worsening | 1 | 2
  Missing | 9 | 4

ADVERSE EVENTS:
Arm/Group | Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 3/136 | 5/135
Other Adverse Events (participants affected / at risk) | 52/136 | 51/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=136) | Placebo (N=135)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Infected bites (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Wound infection pseudomonas (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=136) | Placebo (N=135)
Bronchitis (Infections and infestations) | 7 | 9
Sinusitis (Infections and infestations) | 13 | 9
Upper respiratory tract infection (Infections and infestations) | 15 | 18
Headache (Nervous system disorders) | 7 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 20 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.